CLINICAL TRIAL: NCT02411032
Title: Fresh Start Experiment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Katherine Milkman, Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 820768
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Diabetes; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Reminder control (Experimental): Customers receive a mailing on a random day, which does not coincide with any of the predictable fresh start events.
  Interventions: Behavioral: Reminder
- Birthday framed (Experimental): Customers receive a mailing on the most recent Wednesday before the customers' birthday, and the mailing frames the customers' birthday by emphasizing a fresh start associated with the customers' birthday.
  Interventions: Behavioral: Fresh start; Behavioral: Fresh start framing
- New Year's framed (Experimental): Customers receive a mailing on 1/21/15, and the mailing frames the customers' birthday by emphasizing a fresh start associated with the customers' birthday.
  Interventions: Behavioral: Fresh start; Behavioral: Fresh start framing
- Birthday un-framed (Experimental): Customers receive a mailing on the most recent Wednesday before the customers' birthday, but the mailing does not frame the customers' birthday.
  Interventions: Behavioral: Fresh start
- New Year's un-framed (Experimental): Customers receive a mailing on 1/21/15, but the mailing does not frame New Year's.
  Interventions: Behavioral: Fresh start

INTERVENTIONS:
Behavioral: Reminder — Customer gets mailing that reminds them to take their medication.
  Arms: Reminder control
Behavioral: Fresh start — Customers receive a mailing around a fresh start event: New Year's or birthday
  Arms: Birthday framed; Birthday un-framed; New Year's framed; New Year's un-framed
Behavioral: Fresh start framing — The fresh start event will be highlighted in the mailings.
  Arms: Birthday framed; New Year's framed

SUMMARY:
The investigators are proposing an experiment to help Humana investigate when to launch programs or send messages that are designed to improve customers' engagement. The investigators' past research has shown that certain life events and calendar events (e.g., a job change, a birthday, a holiday, Monday) feel like a "fresh start" to people and have the potential to motivate them to begin pursuing their health goals (e.g., exercising, starting a diet, quitting smoking).

DETAILED DESCRIPTION:
The investigators are proposing an experiment to help Humana investigate when to launch programs or send messages that are designed to improve customers' engagement. The investigators' past research has shown that certain life events and calendar events (e.g., a job change, a birthday, a holiday, Monday) feel like a "fresh start" to people and have the potential to motivate them to begin pursuing their health goals (e.g., exercising, starting a diet, quitting smoking). In this experiment, the investigators will test (a) whether Humana can increase the effectiveness of its messages by sending them to customers around fresh starts moments and (b) whether highlighting a recent fresh start event in Humana's messages can further increase customer engagement.

ELIGIBILITY:
Inclusion Criteria:

* customers of our insurance company partner

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13323 (Actual)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Medication refills | 6 months
  frequency of refilling medication

SECONDARY OUTCOMES:
Hemoglobin A1C | 6 months
LDL cholesterol | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Milkman, Ph.D, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States